CLINICAL TRIAL: NCT02304822
Title: Ciprofloxacin Prophylaxis in Retrograde Intrarenal Surgery: a Prospective Randomized Trail in Comparison of Multiple-, Single- and Zero-dose.
Brief Title: Comparison of Multiple-, Single- and Zero-dose of Ciprofloxacin Prophylaxis in Retrograde Intrarenal Surgery
Acronym: RIRS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guohua Zeng (Other)
Responsible Party: Sponsor-Investigator, Guohua Zeng, Vice-president of The First Affiliated Hospital of Guangzhou Medical University, The First Affiliated Hospital of Guangzhou Medical University
Organization: The First Affiliated Hospital of Guangzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MRER（32）2014
Record Dates: First submitted 2014-11-24; First posted 2014-12-02 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Kidney Stones
Keywords: kidney stones; retrograde intrarenal surgery; ciprofloxacin; prophylaxis; systemic inflammatory response syndrome
MeSH Terms: conditions — Kidney Calculi; Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Multiple-dose of ciprofloxacin prophylaxis (Active Comparator): Multiple-dose prophylactic antibiotic of 200mg intravenous ciprofloxacin, 30 minutes before surgery and within 12 hours after surgery additionally
  Interventions: Drug: Multiple-dose of Ciprofloxacin prophylaxis
- Single-dose of ciprofloxacin prophylaxis (Experimental): Single-dose prophylactic antibiotic of 200mg intravenous ciprofloxacin, 30 minutes before surgery only
  Interventions: Drug: Single-dose of Ciprofloxacin prophylaxis
- Zero-dose of ciprofloxacin prophylaxis (Experimental): Zero-dose of ciprofloxacin prophylaxis with none intravenous ciprofloxacin either preoperatively or postoperatively
  Interventions: Drug: Zero-dose of Ciprofloxacin prophylaxis

INTERVENTIONS:
Drug: Multiple-dose of Ciprofloxacin prophylaxis — Multiple-dose prophylactic antibiotic of 200mg intravenous ciprofloxacin, 30 minutes before surgery and within 12 hours after surgery additionally
  Other Names: Multiple-dose
  Arms: Multiple-dose of ciprofloxacin prophylaxis
Drug: Single-dose of Ciprofloxacin prophylaxis — Single-dose prophylactic antibiotic of 200mg intravenous ciprofloxacin, 30 minutes before surgery only.
  Other Names: Single-dose
  Arms: Single-dose of ciprofloxacin prophylaxis
Drug: Zero-dose of Ciprofloxacin prophylaxis — Zero-dose of ciprofloxacin prophylaxis with none intravenous ciprofloxacin either preoperatively or postoperatively
  Other Names: Zero-dose
  Arms: Zero-dose of ciprofloxacin prophylaxis

SUMMARY:
The purpose of this study is to compare the postoperative systemic inflammatory response syndrome (SIRS) rates undergoing retrograde intrarenal surgery (RIRS) after multiple-, single-, zero-dose of ceftriaxone prophylaxis in a prospective randomized trail.

The investigators will enroll 450 patients who are candidates for RIRS in the investigators study. By simple random sampling technique, patients will be assigned to three groups (multiple-, single-, zero-dose of ceftriaxone prophylaxis,respectively). In addition to the difference of usage of ciprofloxacin prophylaxis, the rest of the procedure is the same in all three groups.The end point of the study is the comparison of outcome of procedure including SIRS rate, stone free rate (SFR), operation time, length of stay,and hematuresis.

DETAILED DESCRIPTION:
PURPOSE:

To compare multiple-, single-, zero-dose antibiotic prophylaxis for retrograde intrarenal surgery (RIRS) and detect the ideal regimen to prevent systemic inflammatory response syndrome (SIRS).

METHODS:

An α error of 5% and a power of 80% were assumed to detect a 14.9% difference in rates of postoperative SIRS (5.1% for the antibiotic prophylaxis group and 20% for the control group) based on the historical data. According to sample size calculation formula for comparing rates between multiple independent samples, n=2λ/(2sin-1√Pmax-2sin-1√Pmin)2,the minimum sample sizes to detect statistically significant differences were estimated to be 86 patients for each of the study groups. To account for patients lost to follow-up and study withdrawals, this number was increased to 100.

After finishing the cases mentioned above, we find the difference in rates of postoperative SIRS in our center is 7.9% (1.2% for the antibiotic prophylaxis group and 9.1% for the control group). According to sample size calculation formula, the minimum sample sizes were estimated to be 124, additional 38 patients are required to be added to each group. For the accuracy and availability of the trial, we decided to enlarge the sample size.To account for patients lost to follow-up and study withdrawals, this number was increased to 150.

After obtaining informed consent, the patients were assessed for eligibility. To allocate the patients, a computer-generated list of random numbers was used. The patients were randomly allocated into three groups by using a randomization ratio of 1:1:1 (group 1, multiple-dose prophylactic antibiotic of 200mg intravenous ciprofloxacin, 30 minutes before surgery and within 12 hours after surgery additionally; group 2, single-dose prophylactic antibiotic of 200mg intravenous ciprofloxacin, 30 minutes before surgery; group 3,zero-dose of prophylactic antibiotic). All patients were operated under intrathecal general anesthesia.

All operations were performed by one experienced surgeon (Guohua Zeng). The surgeon was blinded to group assignment. The postoperative clinical assessment was performed by investigators who had not been involved and were also blind of the group assignment.

Preoperative routine physical examination was performed in all patients. White blood count, blood urea nitrogen, creatinine, liver function test, urinalysis, and urine culture were investigated. Before surgery, stone size and location were determined by choosing at least one of following imaging methods: intravenous pyelography (IVP), kidney, ureter, and bladder (KUB),or unenhanced CT. Inclusion Criteria and exclusion Criteria were shown in the part of "eligibility Criteria".

All equipment used during operation was chosen from the same brand, and standard sterilization procedures were applied. In this study, the investigators used SIRS criteria defined by the committee for consensus on the definition of sepsis, in order to define postoperative fever in a better way. Patients were followed postoperatively according to SIRS criteria: white blood count < 4000 or >12000 cells/mm3, heart rate >90 beats per minute, temperature <36°C or >38°C, respiratory rate > 20 breaths/min. Presence of two or more of these criteria was accepted as SIRS.

RIRS technique :All the endourological procedures in the present study were performed in a standard suite, and a sterile technique was strictly practiced and maintained in all cases. All RIRS procedures were performed under general anesthesia in a low lithotomy position. Ureteroscopy was performed with a semi-rigid 8/9.8Fr ureteroscope (Richard Wolf, Germany), and a flexible 0.035-inch guide wire was inserted into the renal collecting system.A 12/14 Fr ureteral access sheath (Cook Urological, USA) was inserted into the proximal ureter along the guide wire under fluo guiadnce. The Olympus URF-P5 flexible ureteroscope was then advanced via the ureteral access sheath. Irrigation was delivered by manual injection with a 50-mL syringe to achieve a relatively uniform perfusion pressure. Stones were identified and fragmented by holmium: YAG laser lithotripsy. Stone fragments were picked out by the stone basket. Tiny dust and residual fragments < 2 mm were left in place for spontaneous passage. A pigtail 6 Fr Double-J stent was routinely placed at the end of the procedure. The operative time was defined as the time from insertion of an endoscope into the urethra to the completion of stent placement.

Data collection:

Data for the three groups -age, sex, body mass index, laterality of the stone ( left or right), stone surface, stone type (single or multiple), preoperative serum creatinine level, history of hypertension,history of previous surgery, grade of hydronephrosis, operation time, irrigation volume, postoperative serum creatinine level, hemoglobin decrease, duration of hospital stay, initial stone free rate (SFR), final SFR at 1 month, SIRS and hematuresis (modified Clavine system) were recorded.

The stone surface area was measured using computerized systems either on KUB or CT scans. Hospital stay was calculated from operation to discharge from hospital. The operative time was defined as the time from insertion of an endoscope into the urethra to the completion of stent placement. Postoperative SIRS was confirmed by the follow-up 4 weeks after the operation. Stone analysis was performed using infrared spectroscopy. Stone composition was classified according to the European Association of Urology (EAU) guidelines 2015. The JJ stent was removed as an outpatient procedure at 2~4 weeks postoperatively. Postoperative follow-up with a KUB and ultrasound was scheduled at the same time. No observed fragments or fragments smaller than 2 mm was classified as stone free. Complications of all patients were recorded according to the modified Clavien classification system.

The primary endpoints of the study were postoperative SIRS. Secondary endpoints included SFR, operative time, hemoglobin drop and hematuresis.

ELIGIBILITY:
Inclusion Criteria

* Decision to performed RIRS to treat the kidney stones
* American society of Anesthesiology (ASA) score 1 and 2
* Kidney stones of diameter < 2.5 cm

Exclusion Criteria:

* Positive preoperative urine culture
* Pyruria (>10 white blood cells per high-power field)
* Antibiotics treatment of UTI in the last 4 weeks
* Immunocompromised
* Diabetes mellitus
* Allergy to quinolone
* Existing ureteric stents
* Turbid pelvic urine or purulent stone surface observed intraoperatively
* Ureteral stricture, renal or urethral deformity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2014-08 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative SIRS | 4 weeks after RIRS
  White blood count < 4000 or >12000 cells/mm3, heart rate >90 beats per minute, temperature <36°C or >38°C, respiratory rate > 20 breaths/min. Presence of two or more of these criteria was accepted as SIRS.

SECONDARY OUTCOMES:
Stone free rate | 4 weeks after RIRS
  No observed fragments or fragments smaller than 2 mm was classified as stone free.
Hemoglobin drop | Within 24 hours after RIRS
  Hemoglobin drop is assessed by comparing the preoperative hemoglobin level with postoperative hemoglobin level which was detected within 24-hour after RIRS.
Postopeartive hospital stay | During the hospitalization
  Hospital stay was calculated from operation to discharge from hospital.
Operative time | intraoperatively
  The operative time was defined as the time from insertion of an endoscope into the urethra to the completion of stent placement.
Hematuresis | 4 weeks after RIRS
  Macroscopic hematuria was observed.

CONTACTS AND LOCATIONS:
Overall Officials: Guohua Zeng, PH.D and M.D, Study Chair — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Department of Urology, Minimally Invasive Surgery Center, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zhao Z, Fan J, Sun H, Zhong W, Zhu W, Liu Y, Wu W, de la Rosette J, Del Pilar Laguna Pes M, Zeng G. Recommended antibiotic prophylaxis regimen in retrograde intrarenal surgery: evidence from a randomised controlled trial. BJU Int. 2019 Sep;124(3):496-503. doi: 10.1111/bju.14832. Epub 2019 Jun 20. PMID 31136070